CLINICAL TRIAL: NCT01444326
Title: Impact of Dairy Consumption on Inflammation: a Clinical Study
Brief Title: Impact of Dairy Consumption on Inflammation: a Clinical Study (PLI)
Acronym: PLI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Dairy Farmers of Canada (Other)
Responsible Party: Principal Investigator, Benoit Lamarche, Professor, Laval University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: INAF-2010-155
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Cardiovascular Disease
Keywords: Keywords;; Cardiovascular disease; Dairy; Inflammation; Blood lipids
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation | interventions — Dairy Products; Milk; Cheese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dairy diet (Experimental)
  Interventions: Other: Dairy
- Control diet (Placebo Comparator)
  Interventions: Other: Dairy

INTERVENTIONS:
Other: Dairy — During the DAIRY diet, subjects will be asked to incorporate 3 servings of dairy (375 ml of milk, 175 g of yogurt, 30 g of cheese) into their every day diet.
  During the CONTROL arm of the study, participants will be asked to consume energy equivalent replacement products (375 ml of fruit juice, 1 homemade cookie, 20 g of cashew).
  Other Names: Dairy products, milk, cheese, yogourt

SUMMARY:
Inflammation and endothelial dysfunction are being increasingly recognized as key etiological factors in the development of atherosclerosis and subsequent cardiovascular disease (CVD). These pro-atherogenic states are strongly correlated and often found co-segregating among individuals with obesity and the metabolic syndrome. There is increasing evidence to support the use in clinical practice of these novel markers of atherosclerosis and CVD risk. Recent data from the JUPITER study (Justification for the Use of Statins in Primary Prevention: An Intervention Trial Evaluating Rosuvastatin) has provided undisputable evidence that treating patients with elevated plasma CRP concentrations, a marker of systemic subclinical inflammation, leads to marked reduction in the risk of CHD even in patients with highly desirable LDL-C levels. There is also accumulating evidence associating endothelial dysfunction, which is defined as incapacity of the arteries to vasodilate when required, to an increased risk of CVD. While there are more and more studies on how diet affects inflammation and endothelial function, the impact of dairy consumption per se on these novel risk factors for CVD has not been well characterized.

The purpose of this study was to investigate the impact of dairy consumption on markers of inflammation and other risk factors in men and women with low grade systemic inflammation.

DETAILED DESCRIPTION:
This research will be undertaken as a multicenter randomized cross-over controlled study. A total of 140 men and women with subclinical inflammation (plasma CRP 2-10 mg/l) but otherwise healthy will consume two diets, one rich in dairy and one without dairy, while consuming a diet low in saturated fat (<10% energy), in trans fat (<1% energy) and in cholesterol (<200 mg/day). During the DAIRY diet, subjects will be asked to incorporate 3 servings of dairy (milk, yogurt, cheese) into their every day diet. During the CONTROL arm of the study, participants will be asked to consume energy equivalent replacement products. Each diet will be undertaken consecutively in random order and will have duration of approximately 28 days each (4 weeks).The primary analysis consists in comparing inflammation markers and related risk factors between the two treatments. The study is designed to detect a 12-16% difference in plasma CRP concentrations (the primary endpoint) between the control and the dairy diet.

A 2-week stabilization run-in period will precede the randomization of participants. During this run-in period, participants will be asked and instructed to adapt their diet to a prudent dietary pattern low in saturated fat (<10% energy), in trans fat (<1% energy) and in cholesterol (<200 mg/day). The total amount of fat in the diet will not be restricted, with recommendations ranging from 25-35% of energy. However, substitution of saturated for unsaturated fat will be advocated. Sodium intake <2300 mg/d will also be recommended. Recommendations will also include advice on how to restrict the consumption of processed and energy dense foods. The run-in diet will not include specific recommendation on dairy products. Participants will have the choice to include/exclude dairy from their prudent diet, as long as they comply with the main dietary recommendations. This 2-week run-in period will allow participants to familiarize themselves with the dietary recommendations used during the intervention per se. The two diets will be separated by a 4-week wash out period and will also consist to the prudent dietary pattern recommended. It must be stressed that foods will not be provided during the run-in and wash-out periods. These periods are imposed to minimize the inter- and intra-individual variability before and between the experimental phases.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 70 years
* Presenting a subclinical inflammation (Plasma CRP >2 and <10 mg/l)
* Abdominal obesity, waist girth >94 cm in men and >80 cm in women
* Consumption of dairy products fewer than 2 servings per day
* Pre-menopausal women with regular menstrual cycle for the last 3 months

Exclusion Criteria:

* Plasma CRP <2 or >10 mg/l
* Smokers (>1 cigarette/day)
* Body weight variation >10% for the last 6 months prior to the study baseline
* BMI >35 kg/m2
* Previous history of CVD, type 2 diabetes and monogenic dyslipidemia
* Subjects taking medications for hyperlipidemia, hypertension
* Post menopausal women who have initiated hormone replacement therapy within 6 months of study onset
* Endocrine or gastrointestinal disorders
* Smoking
* Food allergies, milk aversion or intolerant to lactose
* Clinical use of vitamin D or calcium supplements
* Vegetarianism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-02 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in plasma CRP concentrations | At the beginning of the study and the end of the two 4-week diets

SECONDARY OUTCOMES:
Change in endothelial function | At the end of the two 4-week diets
Change in plasma lipid concentrations (LDL-Cholesterol, HDL-C, triglycerides) | At the beginning of the study and the end of the two 4-week diets
Change in insulin levels | At the beginning of the study and the end of the two 4-week diets
Change in anthropometric measures (waist and hip circumferences) | At the beginning of the study and the end of the two 4-week diets
Change in blood pressure | At the begining of the study and the end of the two 4-week diets
Change in CRP intravascular kinetics (in a subsample of the entire study population) | At the end of the two 4-week diets

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Lamarche, PhD, Principal Investigator — Laval University
Locations (1):
- Institute of Nutraceutical and Functional Foods (INAF), Laval University, Québec, Quebec, Canada

REFERENCES:
- [Derived] Abdullah MM, Cyr A, Lepine MC, Eck PK, Couture P, Lamarche B, Jones PJ. Common Variants in Cholesterol Synthesis- and Transport-Related Genes Associate with Circulating Cholesterol Responses to Intakes of Conventional Dairy Products in Healthy Individuals. J Nutr. 2016 May;146(5):1008-16. doi: 10.3945/jn.115.222208. Epub 2016 Apr 6. PMID 27052530
- [Derived] Labonte ME, Cyr A, Abdullah MM, Lepine MC, Vohl MC, Jones P, Couture P, Lamarche B. Dairy product consumption has no impact on biomarkers of inflammation among men and women with low-grade systemic inflammation. J Nutr. 2014 Nov;144(11):1760-7. doi: 10.3945/jn.114.200576. Epub 2014 Sep 3. PMID 25332474